CLINICAL TRIAL: NCT04301518
Title: Prematurity Risk Assessment Combined With Clinical Interventions for Improving Neonatal outcoMEs
Acronym: PRIME
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sera Prognostics, Inc. (Industry)
Collaborators: High Risk Pregnancy Center, Las Vegas, Nevada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SP019
Record Dates: First submitted 2020-03-05; First posted 2020-03-10 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Preterm Labor; Preterm Birth
Keywords: neonate; NICU; neonatal; preterm
MeSH Terms: conditions — Obstetric Labor, Premature; Premature Birth

STUDY DESIGN:
Intervention Model Description: To determine the efficacy and safety of a PTB prevention strategy, this study will utilize PreTRM® to prospectively stratify pregnant women with a singleton gestation into categories of risk of PTB and adverse neonatal outcomes. Subjects randomized into the PTB Prevention arm who score at or above the predetermined threshold risk will receive protocol-specified care for the prevention of PTB throughout gestation utilizing defined interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PTB Prevention (Experimental): Approximately 6500 women will be screened, consented, and have the PreTRM® test sample collected. Randomization will occur 1:1 at each site. Those randomized to the PTB Prevention arm will receive the PreTRM® test results. If high risk, women will be consented to take part in the intervention. Those not higher risk will continue on with standard of care.
  Interventions: Other: Multimodal intervention strategy
- Control (No Intervention): Approximately 6500 women will be screened, consented, and have the PreTRM® test sample collected. Randomization will occur 1:1 at each site. Those randomized to the Control arm will not receive the PreTRM® test results. Control arm subjects will continue on with standard of care.

INTERVENTIONS:
Other: Multimodal intervention strategy — * Once weekly nurse support
  * 200 mg/daily micronized progesterone as vaginal suppository
  * 81 mg/daily low dose aspirin
  * two transvaginal ultrasounds
  * cerclage placement if cervical length is less than or equal to 10 mm prior to 24 weeks gestation
  Arms: PTB Prevention

SUMMARY:
This prospective, randomized, controlled study evaluates the safety and efficacy of a preterm birth (PTB) prevention strategy versus standard of care pregnancy management to reduce the incidence of adverse pregnancy outcomes.

DETAILED DESCRIPTION:
Prospective subjects will be randomized to the PTB prevention strategy (PTB Prevention arm) or to standard of care management (Control arm). Subjects randomized to the preterm birth prevention strategy will receive either routine standard of care pregnancy management or a multimodal intervention protocol reserved for higher risk pregnancies based on the results of a commercially-available laboratory developed test, PreTRM® (Sera Prognostics, Inc). The intervention protocol utilizes well-established high-risk pregnancy interventions to improve maternal and neonatal health outcomes.

After enrollment, all subjects will have a blood sample collected once between 18 0/7 weeks and 20 6/7 weeks (126-146 days) of pregnancy. Subjects will be randomized 1:1 to participate in the preterm birth prevention strategy arm or standard of care for pregnancy (Control) arm. Subjects randomized to the Control arm will not receive PreTRM® test results. Subjects randomized to the PTB Prevention arm will receive the results of the PreTRM® test. Results will be reported to the subject, the study Investigator, and the subject's primary pregnancy care provider as "higher risk" of prematurity (≥15%) or "not higher" risk. Subjects with results less than 15% risk (Not Higher Risk Group) by the PreTRM® test will receive standard of care for the duration of pregnancy through hospital discharge. Subjects with results at 15% risk of preterm delivery or greater (Higher Risk Group, equivalent to 2.0-fold the general population risk) by the PreTRM® test will complete a second consenting process to receive a prespecified intervention protocol directed toward reducing risk of adverse pregnancy outcomes inclusive of neonatal morbidity and mortality. All subjects will be followed through the duration of the pregnancy and delivery, and their neonates until initial hospital discharge to assess the course of pregnancy, labor, and any related maternal or fetal complications.

Birth outcomes will be obtained, and liveborn neonates followed through hospital discharge. Readmission of infants will be assessed at 180 days, 1 year and 3 years of life using the HealthCore Integrated Research Database to evaluate longer-term outcomes and costs associated with preterm delivery.

ELIGIBILITY:
Inclusion Criteria

1. Subject is 18 years of age or older
2. Subject is willing and able to provide informed consent and comply with intervention if applicable
3. Subject gestational age is currently within 18 0/7 and 20 6/7 weeks using best estimated due date
4. This is a singleton intrauterine pregnancy
5. Subject has no signs and/or symptoms of preterm labor and has intact membranes
6. Subject has had a 2nd trimester anatomic ultrasound, including evaluation of cervical length, completed by the date of enrollment, but no earlier than 18
7. In the opinion of the Investigator, the subject's delivery data will be accessible within 20 business days from delivery, and neonatal data will be available for data collection purposes within 20 business days from discharge

Exclusion Criteria:

1. Subject has had a prior spontaneous preterm delivery (gestational age at birth less than 37 0/7 weeks gestation)
2. Subject has cervical length less than 25 millimeters (mm) on 2nd trimester transvaginal ultrasound at time of enrollment
3. Subject has taken progesterone or progesterone-derivative medication after 13 6/7 weeks gestation
4. Singleton gestation reduced from an original multiple gestation via embryonic reduction or vanishing twin
5. There is a known major fetal anomaly or chromosomal/ genetic abnormality
6. Placenta accreta spectrum disorder (accreta/ increta/ percreta)
7. Placenta covers the internal os by more than 2.5 centimeters (cm) at time of 2nd trimester anatomic ultrasound (18 0/7 and 20 6/7 weeks gestation)
8. The subject has experienced vaginal bleeding after 13 6/7 weeks gestation
9. One or more of the following uterine risk factors are present: fibroids > 5.0cm, uterine malformation, history of classical cesarean section, history of prior uterine surgery with trans-myometrial penetration (excludes low transverse cesarean section)
10. The subject has a planned cesarean section or induction of labor prior to 370/7 weeks gestation
11. The subject had a cerclage or pessary placed prior to enrollment window in the current pregnancy
12. The subject has received enoxaparin, heparin, heparin sodium or other low molecular weight heparin since last menstrual period
13. Subject has current diagnosis of polyhydramnios
14. Subject has known use of illicit drugs in the current pregnancy, including cocaine, methamphetamine, and/or opioid use disorder in the current pregnancy
15. Subject is allergic to aspirin or has experienced gastrointestinal bleeding associated with use
16. Subject is allergic to peanuts and/or peanut oil used in exogenous progesterone formulation
17. Subject is participating in any other interventional research studies during the current pregnancy
18. Subject has tested positive for COVID-19 via an FDA-authorized diagnostic test for SARS-CoV-2 within the ten days prior to PreTRM® sample collection
19. Subject has been evaluated for COVID-19 salient symptoms per the American College of Obstetrics and Gynecology/ Society for Maternal Fetal Medicine (ACOG/SMFM) "Outpatient Assessment and Management for Pregnant Women with Suspected or Confirmed Novel Coronavirus (COVID-19)" in an emergency room (ER) or hospital setting since the last menstrual period (LMP) date.
20. Subject has a chronic medical disease(s) which require intensive medical surveillance and may increase the risk of preterm delivery to include:

    * Lupus
    * Chronic lung diseases on oxygen replacement
    * Cardiac disease with high risk of maternal mortality, including Marfan syndrome with dilated aortic root and significant pulmonary hypertension
    * Neuromuscular diseases at risk for pulmonary insufficiency (e.g. myotonic dystrophy)
    * Renal failure on dialysis
    * Uncontrolled or poorly controlled hyperthyroidism

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 6500 (Estimated)
Dates: Start 2020-11-06 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Neonatal morbidity/mortality | Through initial neonate discharge from hospital after birth for all neonates, assessed up to 180 days.
  Reduction in composite neonatal morbidity and mortality in the PTB Prevention arm versus the Control arm.
Length of neonatal hospital stay | Through initial neonate discharge from hospital after birth for all neonates, assessed up to 180 days.
  Reduction in length of neonatal hospital stay for admissions from time of birth up to initial neonatal hospital discharge home or neonatal death, whichever occurs first, in the PTB Prevention arm versus the Control arm.

SECONDARY OUTCOMES:
Length of NICU hospital stay for neonates reduction | Through initial neonate discharge from hospital after birth or until neonatal death, whichever occurs first, assessed up to 180 days.
  Reduction in all days spent in the neonatal intensive care unit (NICU) for neonates from time of birth up to discharge home or neonatal death, whichever occurs first, in the PTB Prevention arm versus the Control arm.
Increase gestation | Gestational age at delivery
  Increase in duration of gestation in the PTB Prevention arm versus the Control arm.

OTHER OUTCOMES:
Reduction in occurrence of one or more major neonatal morbidities | 3 year infant follow-up
  Reduction in occurrence of one or more major neonatal morbidities (MNM) with high likelihood of major chronic illness - cystic periventricular leukomalacia, grade 3 and 4 intraventricular hemorrhage, grade 3 or higher retinopathy of prematurity and/or bronchopulmonary dysplasia - in the PTB Prevention arm versus the Control arm.
Cost reduction of neonatal hospitalizations for all admissions | Birth up to neonatal discharge, assessed up to 180 days
  Reduction in all-cause cost of neonatal hospitalizations for all admissions from time of birth up to neonatal discharge in the PTB Prevention arm versus the Control arm in the Anthem beneficiary subset of the study population.
Cost reduction of neonatal hospitalizations for NICU admissions | Birth up to neonatal discharge, assessed up to 180 days
  Reduction in all-cause cost of neonatal hospitalizations, for NICU admissions from time of birth up to neonatal discharge in the PTB Prevention arm versus the Control arm in the Anthem beneficiary subset of the study population.
Cost reduction of neonatal hospitalizations for PTB admissions | Birth up to neonatal discharge, assessed up to 180 days
  Reduction in all-cause cost of neonatal hospitalizations, for PTB admissions from time of birth up to neonatal discharge in the PTB Prevention arm versus the Control arm in the Anthem beneficiary subset of the study population.
Cost reduction of neonatal hospitalizations for PTB admissions after sPTB | Birth up to neonatal discharge, assessed up to 180 days
  Reduction in all-cause cost of neonatal hospitalizations from time of birth up to neonatal discharge for admissions of preterm births after spontaneous rupture of membranes or spontaneous onset of labor (sPTB), in the PTB Prevention arm versus the Control arm in the Anthem beneficiary subset of the study population.
Reduction in rate of preterm birth <32 weeks gestation | Delivery
  Reduction in the rate of preterm birth <32 weeks of gestation in the PTB Prevention arm versus the Control arm.
Reduction in rate of preterm birth <35 weeks gestation | Delivery
  Reduction in the rate of preterm birth <35 weeks of gestation in the PTB Prevention arm versus the Control arm
Reduction in rate of preterm birth <37 weeks gestation | Delivery
  Reduction in the rate of preterm birth <37 weeks of gestation in the PTB Prevention arm versus the Control arm.
Reduction in rate of preterm birth <32 weeks gestation after sPTB | Delivery
  Reduction in the rate of preterm birth <32 weeks of gestation after spontaneous rupture of membranes or spontaneous onset of labor (sPTB), in the PTB Prevention arm versus the Control arm.
Reduction in rate of preterm birth <35 weeks gestation after sPTB | Delivery
  Reduction in the rate of preterm birth <35 weeks of gestation after spontaneous rupture of membranes or spontaneous onset of labor (sPTB), in the PTB Prevention arm versus the Control arm.
Reduction in rate of preterm birth <37 weeks gestation after sPTB | Delivery
  Reduction in the rate of preterm birth <37 weeks of gestation after spontaneous rupture of membranes or spontaneous onset of labor (sPTB), in the PTB Prevention arm versus the Control arm.
NICU days reduction/NICU admissions <37 weeks | Through initial neonatal discharge from hospital after birth or until neonatal death, whichever occurs first, up to 180 days of life
  Reduction in all days spent in the NICU for all NICU admissions of preterm neonates (<37 weeks, only PTB with NICU admission) from birth up to neonatal discharge to home or neonatal death, whichever occurs first, in the PTB Prevention arm versus the Control arm.
NICU days reduction/NICU admissions of sPTB neonates with NICU admission | Through initial neonatal discharge from hospital after birth or until neonatal death, whichever occurs first, up to 180 days of life
  Reduction in all days spent in the NICU for all NICU admissions of spontaneous preterm neonates (only sPTB with NICU admission) from birth up to neonatal discharge to home or neonatal death, whichever occurs first, in the PTB Prevention arm versus the Control arm.
NICU days reduction/NICU admissions of all preterm neonates | Through initial neonatal discharge from hospital after birth or until neonatal death, whichever occurs first, up to 180 days of life
  Reduction in all days spent in the NICU from birth up to neonatal discharge to home or neonatal death, whichever occurs first, for all preterm neonates (independent of NICU admission including zero-length stays for those not admitted), in the PTB Prevention arm versus the Control arm.
NICU days reduction/NICU admissions of sPTB neonates | Through initial neonatal discharge from hospital after birth or until neonatal death, whichever occurs first, up to 180 days of life
  Reduction in all days spent in the NICU from birth up to neonatal discharge to home or neonatal death, whichever occurs first, for all sPTB neonates (independent of NICU admission including zero-length stays for those not admitted), in the PTB Prevention arm versus the Control arm.
Preterm neonatal hospital stay reduction | Through initial neonatal discharge from hospital after birth or until neonatal death, whichever occurs first, up to 180 days of life
  Reduction in length of neonatal hospital stay from birth up to neonatal discharge home or neonatal death, whichever occurs first, for all preterm neonates (<37 weeks, all PTB), in the PTB Prevention arm versus the Control arm.
Preterm neonatal hospital stay reduction for sPTB | Through initial neonatal discharge from hospital after birth or until neonatal death, whichever occurs first, up to 180 days of life
  Reduction in length of neonatal hospital stay from birth up to neonatal discharge home or neonatal death, whichever occurs first, for all preterm neonates (<37 weeks, all sPTB), in the PTB Prevention arm versus the Control arm.
Neonatal hospital and NICU stay reduction after readmission for all admissions | From initial neonatal discharge to home (assessed up to 180 days of life) and within 180 days of life for those discharged prior to 180 days of life
  Reduction in days of total hospital and NICU stay after readmission of infants after initial discharge home and within 180 days of life for all admissions, in the PTB Prevention arm versus the Control arm in the Anthem beneficiary subset of the study population.
Neonatal hospital and NICU stay reduction after readmission for NICU admissions | From initial neonatal discharge to home (assessed up to 180 days of life) and within 180 days of life for those discharged prior to 180 days of life
  Reduction in days of total hospital and NICU stay after readmission of infants after initial discharge home and within 180 days of life for NICU admissions, in the PTB Prevention arm versus the Control arm in the Anthem beneficiary subset of the study population.
Neonatal hospital and NICU stay reduction after readmission for PTB admissions | From initial neonatal discharge to home (assessed up to 180 days of life) and within 180 days of life for those discharged prior to 180 days of life
  Reduction in days of total hospital and NICU stay after readmission of infants after initial discharge home and within 180 days of life for PTB admissions, in the PTB Prevention arm versus the Control arm in the Anthem beneficiary subset of the study population.
Neonatal hospital and NICU stay reduction after readmission for sPTB admissions | From initial neonatal discharge to home (assessed up to 180 days of life) and within 180 days of life for those discharged prior to 180 days of life
  Reduction in days of total hospital and NICU stay after readmission of infants after initial discharge home and within 180 days of life for sPTB admissions, in the PTB Prevention arm versus the Control arm in the Anthem beneficiary subset of the study population.
Hospital readmission cost reduction for all admissions | From initial neonatal discharge to home (assessed up to 180 days of life) and within 180 days of life for those discharged prior to 180 days of life
  Reduction in all-cause costs of hospital readmission of infants after initial discharge and within 180 days of life for all admissions, in the PTB Prevention arm versus the Control arm in the Anthem beneficiary subset of the study population.
Hospital readmission cost reduction for NICU admissions | From initial neonatal discharge to home (assessed up to 180 days of life) and within 180 days of life for those discharged prior to 180 days of life
  Reduction in all-cause costs of hospital readmission of infants after initial discharge and within 180 days of life for NICU admissions, in the PTB Prevention arm versus the Control arm in the Anthem beneficiary subset of the study population.
Hospital readmission cost reduction for PTB admissions | From initial neonatal discharge to home (assessed up to 180 days of life) and within 180 days of life for those discharged prior to 180 days of life
  Reduction in all-cause costs of hospital readmission of infants after initial discharge and within 180 days of life for PTB admissions, in the PTB Prevention arm versus the Control arm in the Anthem beneficiary subset of the study population.
Hospital readmission cost reduction for sPTB admissions | From initial neonatal discharge to home (assessed up to 180 days of life) and within 180 days of life for those discharged prior to 180 days of life
  Reduction in all-cause costs of hospital readmission of infants after initial discharge and within 180 days of life for sPTB admissions, in the PTB Prevention arm versus the Control arm in the Anthem beneficiary subset of the study population.
Hospital readmission cost reduction for all admissions within first year of life | From initial neonatal discharge to home (assessed up to 180 days of life) and within first year of life
  Reduction in all-cause costs of hospital readmission of infants after initial discharge and within the first year of life for all admissions, in the PTB Prevention arm versus the Control arm in the Anthem beneficiary subset of the study population.
Hospital readmission cost reduction within first year of life for NICU admissions | From initial neonatal discharge to home (assessed up to 180 days of life) and within first year of life
  Reduction in all-cause costs of hospital readmission of infants after initial discharge and within the first year of life for NICU admissions, in the PTB Prevention arm versus the Control arm in the Anthem beneficiary subset of the study population.
Hospital readmission cost reduction within first year of life for PTB admissions | From initial neonatal discharge to home (assessed up to 180 days of life) and within first year of life
  Reduction in all-cause costs of hospital readmission of infants after initial discharge and within the first year of life for PTB admissions, in the PTB Prevention arm versus the Control arm in the Anthem beneficiary subset of the study population.
Hospital readmission cost reduction within first year of life for sPTB admissions | From initial neonatal discharge to home (assessed up to 180 days of life) and within first year of life
  Reduction in all-cause costs of hospital readmission of infants after initial discharge and within the first year of life for sPTB admissions, in the PTB Prevention arm versus the Control arm in the Anthem beneficiary subset of the study population.
Hospital readmission cost reduction within first three years of life for all admissions | From initial neonatal discharge to home (assessed up to 180 days of life) and within first three years of life
  Reduction in all-cause costs of hospital readmission of infants after initial discharge and within the first three years of life for all admissions, in the PTB Prevention arm versus the Control arm in the Anthem beneficiary subset of the study population.
Hospital readmission cost reduction within first three years of life for NICU admissions | From initial neonatal discharge to home (assessed up to 180 days of life) and within first three years of life
  Reduction in all-cause costs of hospital readmission of infants after initial discharge and within the first three years of life for NICU admissions, in the PTB Prevention arm versus the Control arm in the Anthem beneficiary subset of the study population.
Hospital readmission cost reduction within first three years of life for PTB admissions | From initial neonatal discharge to home (assessed up to 180 days of life) and within first three years of life
  Reduction in all-cause costs of hospital readmission of infants after initial discharge and within the first three years of life for PTB admissions, in the PTB Prevention arm versus the Control arm in the Anthem beneficiary subset of the study population.
Hospital readmission cost reduction within first three years of life for sPTB admissions | From initial neonatal discharge to home (assessed up to 180 days of life) and within first three years of life
  Reduction in all-cause costs of hospital readmission of infants after initial discharge and within the first three years of life for sPTB admissions, in the PTB Prevention arm versus the Control arm in the Anthem beneficiary subset of the study population.
NICU admission rate reduction | Through initial neonatal discharge from hospital after birth or until neonatal death, whichever occurs first, assessed up to 180 days
  Reduction in NICU admission rates in the immediate neonatal period prior to initial discharge home or neonatal death, whichever occurs first, in the PTB Prevention arm versus Control arm.
Neonatal morbidity and mortality index observation | Within one year of primary analysis
  Observation of the dependence of the composite neonatal morbidity and mortality index co-primary endpoint on severity of risk as defined by PreTRM® categorical test results and continuous risk score, both in comparison of the PTB Prevention arm versus the Control arm and with stratification of both arms by PreTRM® test result.
Neonatal hospital length of stay observation | Within one year of primary analysis
  Observation of the dependence of the length of neonatal hospital stay co-primary endpoint on severity of risk as defined by PreTRM® categorical test results and continuous risk score, both in comparison of the PTB Prevention arm versus the Control arm and with stratification of both arms by PreTRM® test result.
NICU length of stay observation | Within one year of primary analysis
  Observation of the dependence of the NICU length of stay secondary endpoint on severity of risk as defined by PreTRM® categorical test results and continuous risk score, both in comparison of the PTB Prevention arm versus the Control arm and with stratification of both arms by PreTRM® test result.
Duration of gestation observation | Within one year of primary analysis
  Observation of the dependence of the duration of gestation secondary endpoint on severity of risk as defined by PreTRM® categorical test results and continuous risk score, both in comparison of the PTB Prevention arm versus the Control arm and with stratification of both arms by PreTRM® test result.
Major neonatal morbidities observation | Within one year of primary analysis
  Observation of the dependence of the MNM exploratory endpoint on severity of risk as defined by PreTRM® categorical test results and continuous risk score, both in comparison of the PTB Prevention arm versus the Control arm and with stratification of both arms by PreTRM® test result.
NICU length of stay amongst preterm neonates observation | Within one year of primary analysis
  Observation of the dependence of the exploratory endpoint of dependence of NICU length of stay amongst preterm neonates on severity of risk as defined by PreTRM® categorical test results and continuous risk score, both in comparison of the PTB Prevention arm versus the Control arm and with stratification of both arms by PreTRM® test result.
Hospital length of stay amongst preterm neonates observation | Within one year of primary analysis
  Observation of the dependence of the exploratory endpoint of dependence of hospital length of stay amongst preterm neonates on severity of risk as defined by PreTRM® categorical test results and continuous risk score, both in comparison of the PTB Prevention arm versus the Control arm and with stratification of both arms by PreTRM® test result.
Preterm birth rate observation | Within one year of primary analysis
  Observation of the dependence of the preterm birth rate exploratory endpoint on severity of risk as defined by PreTRM® categorical test results and continuous risk score, both in comparison of the PTB Prevention arm versus the Control arm and with stratification of both arms by PreTRM® test result.
Neonatal hospitalization cost observation | Within one year of primary analysis
  Observation of the dependence of the exploratory endpoint of all-cause cost of neonatal hospitalization on severity of risk as defined by PreTRM® categorical test results and continuous risk score, both in comparison of the PTB Prevention arm versus the Control arm and with stratification of both arms by PreTRM® test result.
Preterm neonatal hospitalization observation | Within one year of primary analysis
  Observation of the dependence of the exploratory endpoint of all-cause cost of neonatal hospitalization amongst preterm neonates on severity of risk as defined by PreTRM® categorical test results and continuous risk score, both in comparison of the PTB Prevention arm versus the Control arm and with stratification of both arms by PreTRM® test result.
Intervention protocol observation/neonatal morbidity and mortality index | Within one year of primary analysis
  Observation of the contribution of components of the intervention protocol, including consideration of consent and adherence, to the co-primary endpoint of composite neonatal morbidity and mortality index.
Intervention protocol observation/length of neonatal hospital stay | Within one year of primary analysis
  Observation of the contribution of components of the intervention protocol, including consideration of consent and adherence, to the co-primary endpoint of length of neonatal hospital stay.
Intervention protocol observation/length of NICU stay | Within one year of primary analysis
  Observation of the contribution of components of the intervention protocol, including consideration of consent and adherence, to the, secondary endpoint of length of NICU stay.
Intervention protocol observation/duration of gestation | Within one year of primary analysis
  Observation of the contribution of components of the intervention protocol, including consideration of consent and adherence, to the secondary endpoint of duration of gestation.
Intervention protocol observation/major neonatal morbidities | Within one year of primary analysis
  Observation of the contribution of components of the intervention protocol, including consideration of consent and adherence, to the MNM and exploratory endpoint.
Intervention protocol observation/length of NICU stay amongst preterm neonates | Within one year of primary analysis
  Observation of the contribution of components of the intervention protocol, including consideration of consent and adherence, to the exploratory endpoint of length of NICU stay amongst preterm neonates.
Intervention protocol observation/length of hospital stay amongst preterm neonates | Within one year of primary analysis
  Observation of the contribution of components of the intervention protocol, including consideration of consent and adherence, to the exploratory endpoint of length of hospital stay amongst preterm neonates.
Intervention protocol observation/preterm birth rate | Within one year of primary analysis
  Observation of the contribution of components of the intervention protocol, including consideration of consent and adherence, to the exploratory endpoint of preterm birth rate.
Intervention protocol observation/neonatal hospitalization | Within one year of primary analysis
  Observation of the contribution of components of the intervention protocol, including consideration of consent and adherence, to the exploratory endpoint of all-cause cost of neonatal hospitalization.
Intervention protocol observation/neonatal hospitalization amongst preterm neonates | Within one year of primary analysis
  Observation of the contribution of components of the intervention protocol, including consideration of consent and adherence, to the exploratory endpoint of all-cause cost of neonatal hospitalization amongst preterm neonates.
COVID-19 primary | Within one year of primary analysis
  Observation of the effect on primary endpoints of SARS-CoV-2 positivity or COVID-19 salient symptoms requiring evaluation in an ER or hospital setting after enrollment.
COVID-19 secondary | Within one year of primary analysis
  Observation of the effect on secondary endpoints of SARS-CoV-2 positivity or COVID-19 salient symptoms requiring evaluation in an ER or hospital setting after enrollment.
COVID-19 exploratory | Within one year of primary analysis
  Observation of the effect on exploratory endpoints of SARS-CoV-2 positivity or COVID-19 salient symptoms requiring evaluation in an ER or hospital setting after enrollment.
Anxiety - Generalized Anxiety Disorder 7-item (GAD-7) | Within one year of primary analysis
  Change (mean difference) in Generalized Anxiety Disorder 7-item (GAD-7) scores at enrollment and 6-weeks post-enrollment in a subset of subjects. Scale range 0 - 21, higher values correlate with higher anxiety
Anxiety - Perinatal Anxiety Screening Scale (PASS) | Within one year of primary analysis
  Change (mean difference) in perinatal Anxiety Screening Scale (PASS) scores at enrollment and 6-weeks post-enrollment in a subset of subjects. Scale range 0 - 93, higher values correlate with higher anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Brian Iriye, MD, Principal Investigator — High Risk Pregnancy Center
Locations (18):
- United States (18):
  - UCSD, San Diego, California
  - Yale, New Haven, Connecticut
  - Delaware/Christiana Care, Newark, Delaware
  - Emerald Coast, Panama City, Florida
  - University of Kentucky Healthcare, Lexington, Kentucky
  - Ochsner, New Orleans, Louisiana
  - LSU, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Beaumont Hospital, Royal Oak, Michigan
  - High Risk Pregnancy Center, Las Vegas, Nevada
  - Mt Sinai, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio Health, Columbus, Ohio
  - UTMB, Galveston, Texas
  - University of Virginia, Charlottesville, Virginia
  - Inova Health Care Services, Falls Church, Virginia
  - VPFW, Richmond, Virginia
  - MCW, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No